CLINICAL TRIAL: NCT07086768
Title: A Phase Ia/Ib, 2-Part, Dose-Escalation and Dose-Expansion Study of BSI-082 Monotherapy and Combined Therapy in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Dose-Escalation and Dose-Expansion Study of BSI-082 Monotherapy and Combined Therapy in Patients With Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lei Zheng (Other)
Collaborators: Biosin USA, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Lei Zheng, Executive Director of University of Texas Health Science Center at San Antonio Cancer Center, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 25-0042
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: anti-SIRPα antibody; anti-signal regulatory protein alpha; Dose Escalation; Dose Expansion
MeSH Terms: conditions — Neoplasm Metastasis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: This is a phase Ia/Ib, open-label, dose-escalation and dose-expansion study designed to evaluate BSI-082 monotherapy and combined therapy with Trastuzumab deruxtecan (T-DXd) in patients with locally advanced or metastatic solid tumors.
  A Phase 1a/1b, open-label, dose-escalation and dose expansion study. This study will have 2 parts: Phase Ia monotherapy dose-escalation and Phase Ib combination and dose-expansion.A traditional 3+3 method will be applied for dose escalation phase for Phase 1a. Phase 1b will have 2 dose cohorts, a lower dose and a higher dose cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: monotherapy (Experimental): BSI-082 0.3mg/kg will be administrated as an IV infusion on Day 1 of each 21-day treatment cycle
  Interventions: Drug: BSI-082
- Cohort 2: monotherapy (Experimental): BSI-082 1mg/kg will be administrated as an IV infusion on Day 1 of each 21-day treatment cycle
  Interventions: Drug: BSI-082
- Cohort 3: monotherapy (Experimental): BSI-082 3mg/kg will be administrated as an IV infusion on Day 1 of each 21-day treatment cycle
  Interventions: Drug: BSI-082
- Cohort 4: monotherapy (Experimental): BSI-082 10mg/kg will be administrated as an IV infusion on Day 1 of each 21-day treatment cycle
  Interventions: Drug: BSI-082
- Cohort 5: monotherapy (Experimental): BSI-082 20mg/kg will be administrated as an IV infusion on Day 1 of each 21-day treatment cycle
  Interventions: Drug: BSI-082
- Cohort b1: combined therapy (Experimental): Lower dose cohort of BSI-082 with established dose of T-DXd
  Interventions: Drug: BSI-082; Other: Trastuzumab deruxtecan
- Cohort b2: combined therapy (Experimental): Higher dose cohort of BSI-082 with established dose of T-DXd
  Interventions: Drug: BSI-082; Other: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: BSI-082 — BSI-082 is a sterile solution for injection which contains the active ingredient at the nominal concentration of 50.0 mg/mL. T
Other: Trastuzumab deruxtecan — T-DXd: Administrate as per the drug package insert and Investigator's guidance, and T-DXd can be continued after the patients been taken off from the study.
  Other Names: Standard of care treatment with
  Arms: Cohort b1: combined therapy; Cohort b2: combined therapy

SUMMARY:
This is a study that will enroll patients with cancer who have tumors that may have spread. The patients will know what medication they are being given.

There will be 2 parts to the study. For the first part of the study only one medication will be taken, and the dose changed to a higher dose over time.

In the second part of the study tow medications will be taken and the dose of the medication may be changed to a higher dose.

DETAILED DESCRIPTION:
Phase 1a monotherapy dose-escalation part will establish the safety and tolerability of BSI-082 as single agent. Up to 30 patients with locally advanced or metastatic solid tumors who have relapsed, or been non-responsive, or have developed disease progression through standard systemic therapy, or have been ineligible for standard systemic therapy known to confer clinical benefit will be enrolled. Recommended dose for expansion (RDE) will be determined in this phase and used in the phase 1b study.

Phase 1b combination dose-escalation and dose-expansion part will enroll up to 27 patients with Her2 positive locally advanced solid tumors that are indicated for the Standard of care T-DXd treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Read, understood, and provided written informed consent and must be willing to comply with all study requirements and procedures.
2. Adults ≥ 18 years of age at the time of informed consent form is signed.
3. Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors who have relapsed, or been non-responsive, or have developed disease progression through standard systemic therapy, or have been ineligible for standard systemic therapy known to confer clinical benefit.
4. Patients having an FDA-approved indication for T-DXd (only for Phase 1b dose expansion).
5. With 4 weeks or 5 half-lives (whichever is shorter) of prior anticancer therapies (only for Phase 1a dose escalation).
6. Life expectancy ≥ 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
8. Presence of at least 1 measurable lesion based on computed tomography (CT) or magnetic resonance imaging (MRI) per RECISIT V1.1.
9. Has a left ventricular ejection fraction (LVEF) ≥50% by either an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before enrollment.
10. Main organ functions meet the following criteria:

    * Absolute Neutrophil Count (ANC) ≥ 1.5×109/L
    * Platelet counts ≥ 100×109/L
    * Hemoglobin ≥ 9 g/dL (without recent red blood cell transfusion within 2 weeks prior to study entry)
    * Creatinine clearance ≥ 40 mL/min per the Cockcroft and Gault formula.
    * AST ≤ 2.5×Upper Limit Normal (ULN or patients with hepatic metastasis ≤ 5×ULN
    * ALT ≤ 2.5×ULN or patients with hepatic metastasis ≤ 5×ULN
    * Total Bilirubin ≤ 1.5×ULN, except for patients with Gilbert's syndrome from whom total bilirubin < 3.0 × ULN or direct bilirubin < 1.5 × ULN
11. Both male and female of childbearing potential patients enrolled in this trial as well as their partners must agree to use highly effective contraception during the study and for at least 10 months after discontinuing study treatment. Patients and/or partners who are surgically sterile or postmenopausal are exempt from this requirement.

Exclusion Criteria:

1. Known allergies, hypersensitivity, or intolerance to monoclonal antibodies (mAbs) or formulation components of BSI-082.
2. Prior therapy with any SIRPα or CD47 targeting agents.
3. Has active autoimmune disease or a documented history of autoimmune disease, or history of potential autoimmune syndrome that required systemic steroids or immunosuppressive medications, except for patients with vitiligo, endocrinopathies, type 1 diabetes, or patients with resolved childhood asthma/atopy or other syndromes which would not be expected to recur in the absence of an external trigger (e.g., drug-related serum sickness or post-streptococcal glomerulonephritis). Patients with mild asthma who require intermittent use of bronchodilators (such as albuterol) and those who have not been hospitalized for asthma in the preceding 3 years will not be excluded from this study.
4. Toxicities of prior anticancer therapies have not resolved to ≤ Grade 1 or to baseline) prior to the first dose of study treatment (excluding alopecia, vitiligo, endocrinopathies on stable hormone replacement therapy, Grade 2 neuropathy from taxanes or platinum containing therapies and Grade 2 hearing loss from platinum-containing therapies).
5. Has other malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers; or any other cancer from which the patient has been disease-free for at least 5 years.
6. Occurrence of immune related toxicity necessitating permanent discontinuation or immune related toxicity that required treatment with a TNF inhibitor (e.g., infliximab) in patients with previous immunotherapy.
7. Medical history of myocardial (MI) within 6 months before study enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Class II to IV).
8. Any of the following within 6 months of enrollment: cerebrovascular accident, transient ischemic attack, other arterial thromboembolic events, or pulmonary embolism.
9. Has a QT interval corrected with Fridericia's formula (QTcF) prolongation to >470 ms based on average of the screening triplicate 12-lead electrocardiogram (ECG).
10. Uncontrolled hypertension (resting systolic blood pressure>180 mmHg or diastolic blood pressure>110 mmHg) and/or severe arrhythmia within 28 days before enrollment.
11. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
12. Has lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder.
13. Any autoimmune, connective tissue or inflammatory disorders where there is documented or suspicion of pulmonary involvement at the time of screening.
14. Prior complete pneumonectomy.
15. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
16. Has uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals.
17. Has active primary immunodeficiency or active human immunodeficiency virus (HIV) infection as determined by plasma HIV ribonucleic acid (RNA) viral load and CD4 count. For the Dose-expansion phase only, participants with undetectable viral load or normalized CD4 count (CD4+ T-cell counts ≥ 350 cells/μL) and no opportunistic infection within the past 12 months will be eligible. These participants must be on established antiretroviral therapy for at least 4 weeks and have an HIV viral load <400 copies/mL prior to enrollment.
18. Has active hepatitis B or C infection. Participants with past hepatitis C virus (HCV) infection and positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA. Participants with past or resolved hepatitis B virus infection are eligible only if confirmed by the Investigator.
19. Has received a live, attenuated vaccine (messenger ribonucleic acid [mRNA] and replication-deficient adenoviral vaccines are not considered live, attenuated vaccines) within 30 days prior to first exposure to study drug(s).
20. Has any other acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results would make the patient inappropriate for entry into the trial.
21. Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may interfere with the participant's participation in the clinical study or evaluation of the clinical study results.
22. Women who are pregnant or lactating. All female patients of childbearing potential must have a negative serum pregnancy test prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-07 (Estimated); Study Completion 2028-08-07 (Estimated)

PRIMARY OUTCOMES:
Number of Dose limiting toxicity Events | Baseline to 42 days
  Adverse events (AEs) as characterized by type, frequency, severity (as graded by national cancer institute common terminology criteria for adverse events, NCI CTCAE V5.0), timing, seriousness, and relationship to study treatment.
  •And Vital sign abnormalities and laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE V5.0) and timing.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, MD, Study Director — The University of Texas Health Science Center at San Antonio; John Sarantopoulos, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio

IPD SHARING:
Plan to Share IPD: Yes
Any manuscript, abstract or other publication or presentation of results or information arising in connection with the trial (including any ancillary trial involving trial subjects) must be prepared in conjunction with the Mays Cancer Center Data Safety Monitoring Board, the trial's statistician, and verification that all study data to be used for the publication has been monitored for accuracy by the Mays Quality Assurance (QA) team prior to publication or presentation.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion and data analysis for publication.